CLINICAL TRIAL: NCT04835129
Title: A Multisite, Phase II Study of Isatuximab, Pomalidomide, Elotuzumab and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Brief Title: Isatuximab, Pomalidomide, Elotuzumab and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Acronym: IMPEDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00041365
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: relapsed and/or refractory multiple myeloma; salvage therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; pomalidomide; elotuzumab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety Run-in (Experimental): Six subjects will be enrolled. Isatuximab (10 mg/kg) intravenous (IV) on days 2, 8, 15, 22 of cycle 2 and days 1 and 15 of subsequent cycles. Pomalidomide (4 mg) by mouth (PO) days 1-21 of each cycle. Elotuzumab (10 mg/kg) on days 1, 8, 15, 22 of cycles 1 and 2; 20 mg/kg on day 1 of subsequent cycles. Dexamethasone 40 mg (20 mg if >75 years) PO or IV on days 1, 8,15 and 22 of each cycle.
  Interventions: Drug: Isatuximab (for run-in portion); Drug: Pomalidomide; Drug: Elotuzumab; Drug: Dexamethasone
- Expansion (Experimental): Forty-seven subjects with relapsed and/or refractory multiple myeloma will be enrolled.
  Isatuximab (10 mg/kg) IV on days 2, 8, 15, 22 of cycle 1 and days 1 and 15 of subsequent cycles. Pomalidomide (4 mg) PO days 1-21 of each cycle. Elotuzumab (10 mg/kg) on days 1, 8, 15, 22 of cycles 1 and 2; 20 mg/kg on day 1 of subsequent cycles. Dexamethasone 40 mg (20 mg if >75 years) PO or IV on days 1, 8,15 and 22 of each cycle.
  Interventions: Drug: Isatuximab (for expansion); Drug: Pomalidomide; Drug: Elotuzumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab (for run-in portion) — 10 mg/kg IV on days 2, 8, 15, 22 of cycle 2 and days 1 and 15 of subsequent cycles.
  Other Names: Sarclisa; SAR-650984; isatuximab-irfc
  Arms: Safety Run-in
Drug: Isatuximab (for expansion) — 10 mg/kg IV on days 2, 8, 15, 22 of cycle 1 and days 1 and 15 of subsequent cycles.
  Other Names: Sarclisa; SAR-650984; isatuximab-irfc
  Arms: Expansion
Drug: Pomalidomide — 4 mg PO days 1-21 of each cycle.
  Other Names: Pomalyst; Imnovid
Drug: Elotuzumab — 10 mg/kg on days 1, 8, 15, 22 of cycles 1 and 2; 20 mg/kg on day 1 of subsequent cycles.
  Other Names: Empliciti; HuLuc63
Drug: Dexamethasone — 40 mg (20 mg if >75 years) PO or IV on days 1, 8,15 and 22 of each cycle.
  Other Names: Baycadron; Decadron; DexPak; TaperDex; Zema-Pak; ZoDex; Zonacort

SUMMARY:
This is a multicenter, open-label phase II study in subjects with relapsed and/or refractory multiple myeloma with at least two prior lines of therapy. The main study consists of three phases: a 28-day screening phase, treatment phase that consists of 28-day cycles of isatuximab with elotuzumab, pomalidomide, and dexamethasone and a follow-up phase.

DETAILED DESCRIPTION:
The study is divided into two parts:

Part 1 (Run-in safety phase): In this safety-run in phase a total of six subjects will be enrolled at the coordinating site (Medical College of Wisconsin) to assess potential dose-limiting toxicities that may be associated with the addition of isatuximab with pomalidomide, elotuzumab and dexamethasone.

Part 2 (Expansion phase): In this part, up to 47 additional subjects will be enrolled.

The study hypothesis is that the isatuximab in combination with elotuzumab, pomalidomide, and dexamethasone (Isa-EPD) will be safe and lead to superior response rates than seen with either isatuximab with pomalidomide and dexamethasone or elotuzumab with pomalidomide and dexamethasone in subjects with relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent must be given before performance of any study related procedure.
2. Male or female subjects ≥18 years.
3. Multiple myeloma subjects with at least 2 prior therapies that included lenalidomide and proteasome inhibitor combined or in different regimens, and refractory to most recent line of therapy.
4. Measurable disease as defined by any of the following:

   * Serum M-protein level ≥0.5 g/dL OR
   * Urine M-protein level ≥200 mg/24 hours; OR
   * Light chain multiple myeloma without measurable disease in the urine: serum Ig free light chains (FLC) ≥10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Female subjects who:

   1. Are postmenopausal (see Appendix 4 for definition) for at least one year before the screening visit, OR
   2. Are surgically sterile, OR
   3. Females of childbearing potential or male subjects with female partners of childbearing potential shall be required to use effective contraceptive methods (double barrier method, intrauterine device, oral contraception or abstinence) starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s). A woman is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Any of the following highly effective methods of contraception are accepted:

      * Established use of oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation.
      * Established use of oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation.
      * Placement of an intrauterine device or intrauterine hormone-releasing system.
      * Barrier methods of contraception: male condom with either cap, diaphragm or sponge with spermicide (double-barrier methods). The use of double-barrier methods should always be supplemented with the use of a spermicide. Female condom and male condom should not be used together.
      * Male sterilization (provided that the partner is the sole sexual partner of the subject and that the sterilized partner has received medical assessment of the surgical success).
      * Sexual abstinence.
      * Female subjects must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
   4. Females of childbearing potential must have a negative serum or urine pregnancy test prior to enrollment.
7. Male subjects, even if surgically sterilized (i.e., status post vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through four months after the last dose of study drug(s) (female and male condoms should not be used together), or
   2. Agree to practice true abstinence during the entire study treatment period from the time of signing the informed consent through four months after the last dose of study drug(s), when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
8. Due to the teratogenicity of pomalidomide and the lack of adequate reproductive toxicity data for isatuximab and/or elotuzumab, in addition to the user independent highly effective method of contraception, a male or female condom with or without spermicide, diaphragm, or cervical cap is required. Male condom and female condom should not be used together (due to risk of failure with friction).

Exclusion Criteria:

1. Diagnosed or treated for malignancy other than multiple myeloma, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥3 years before enrollment.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ (e.g., cervical, breast) with no evidence of disease.
2. Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma.
3. Subjects refractory to prior signaling lymphocytic activation molecule F7 (SLAMF7) monoclonal antibody
4. Prior cluster of differentiation 38 (CD38) monoclonal antibody is allowed as long it has been >6 months and patients had achieved at least a partial response or better.
5. Subject refractory or intolerant to prior pomalidomide therapy.
6. Known chronic obstructive pulmonary disease
7. Known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. Note: Subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study.
8. Known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have untreated or active hepatitis C.
9. Concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
10. Clinically significant cardiac disease, including:

    * Myocardial infarction within six months before enrollment or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
    * Uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] Version 5 Grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
    * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
    * Uncontrolled hypertension (BP >160/100 in the presence of blood pressure medications)
11. Subjects who have inadequate evidence of bone marrow/hepatic/renal function as defined by the following:

    * Absolute neutrophil count <1.0 × 109/L; no growth factors in the previous seven days is allowed.
    * Hemoglobin level ≤7.5 g/dL (≤5 mmol/L); blood transfusions to maintain hemoglobin >7.5 g/dL are acceptable.
    * Platelet count <75 × 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise, platelet count <50 × 109/L; no platelet transfusions in the past seven days are allowed.
    * Alanine aminotransferase (ALT) level ≥2.5 × ULN
    * Aspartate aminotransferase (AST) level ≥2.5 × ULN
    * Total bilirubin level ≥1.5 × ULN, (except for Gilbert Syndrome: direct bilirubin ≥2 × ULN)
    * Corrected serum calcium >14.0 mg/dL (>3.5 mmol/L) or free ionized calcium >6.5 mg/dL (>1.6 mmol/L)
12. Known allergies, hypersensitivity (if not amenable to premedication with steroids, or H2 blockers), or intolerance to monoclonal antibodies or human proteins, isatuximab or its excipients or known sensitivity to mammalian-derived products.
13. Plasma cell leukemia (>2.0 × 10^9/L circulating plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and/or skin changes), or light-chain amyloidosis.
14. Known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
15. Pregnant or breastfeeding or planning to become pregnant starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
16. Plans to father a child starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
17. Had major surgery within two weeks before Cycle 1, Day 1, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within two weeks after the last dose of study drug administration. Note: Subjects with planned surgical procedures to be conducted under local anesthesia are not excluded. Kyphoplasty is not considered a major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects in each status category of the International Myeloma Working Group (stringent complete response, complete response, very good partial response, partial response, minimal response, stable disease, progressive disease). | Year 1
  This will be measured using the International Myeloma Working Group criteria. For clarity, the response will be reported at the end of each treatment year.
The number of subjects in each status category of the International Myeloma Working Group (stringent complete response, complete response, very good partial response, partial response, minimal response, stable disease, progressive disease). | Year 2
  This will be measured using the International Myeloma Working Group criteria. For clarity, the response will be reported at the end of each treatment year.
The number of subjects in each status category of the International Myeloma Working Group (stringent complete response, complete response, very good partial response, partial response, minimal response, stable disease, progressive disease). | Year 3
  This will be measured using the International Myeloma Working Group criteria. For clarity, the response will be reported at the end of each treatment year.

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158